CLINICAL TRIAL: NCT03779230
Title: A Study to Evaluate the Safety and Efficacy of the Tumor-targeting Human Antibody-cytokine Fusion Protein L19TNF in Patients With Isocitrate Dehydrogenase (IDH) Wildtype WHO Grade III / IV Glioma at First Relapse
Brief Title: Safety and Efficacy of L19TNF in Patients With Isocitrate Dehydrogenase (IDH) Wildtype WHO Grade III / IV Glioma at First Relapse
Acronym: GLIOMOON
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19TNFGLIO-02/18
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Glioma of Brain

STUDY DESIGN:
Intervention Model Description: Open label, non-randomized, mono-center Phase I/II study in subjects with IDH-wildtype WHO grade III / IV glioma at first relapse.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- L19TNF (Experimental): Patients will be assigned to the following increasing dose levels of L19TNF: 10 and 13 μg/kg.
  Interventions: Drug: L19TNF

INTERVENTIONS:
Drug: L19TNF — Patients will be assigned to the following increasing dose levels of L19TNF: 10 and 13 μg/kg.
  Other Names: onfekafusp alpha

SUMMARY:
Open label, non-randomized, mono-center Phase I/II study in subjects with IDH-wildtype WHO grade III / IV glioma at first relapse.

DETAILED DESCRIPTION:
The purpose of this study is to explore the safety and efficacy profile of the antibody-cytokine fusion protein L19TNF in patients with isocitrate dehydrogenase (IDH) wildtype WHO grade III / IV glioma at first relapse

Phase I:

The primary objective of this phase is to evaluate the safety of L19TNF in patients with IDH-wildtype WHO grade III / IV glioma at first relapse and to establish and confirm the recommended dose (RD) for phase II.

Phase II:

The primary objective of this phase is to evaluate antitumor activity of L19TNF in patients with IDH-wildtype WHO grade III / IV glioma at first relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 or more
2. Patients with histologically confirmed IDH-wildtype WHO grade III / IV glioma at first relapse
3. Radiographic demonstration of disease progression
4. Presence of at least one lesion of bi-dimensionally measurable disease by MRI of at least 1 cm (10 mm) in the longest diameter on baseline MRI.
5. Karnofsky Performance Score (KPS) ≥ 70%
6. Documented negative test for HIV-HBV-HCV. For HBV serology: the determination of HBsAg, anti-HBsAg-Ab and anti-HBcAg-Ab is required. In patients with serology documenting previous exposure to HBV (i.e., anti-HBs Ab with no history of vaccination and/or anti-HBc Ab), negative serum HBV-DNA is required. For HCV: HCV-RNA or HCV antibody test. Subjects with a positive test for HCV antibody but no detection of HCV-RNA indicating no current infection are eligible.
7. Female patients: negative pregnancy test for women of childbearing potential (WOCBP)* within 14 days of starting treatment. WOCBP must agree to use, from the screening to six months following the last study drug administration, highly effective contraception methods, as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group (www.hma.eu/ctfg.html) and which include, for instance, progesteron-only or combined (estrogen- and progesteron-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion or vasectomized partner.

   Male patients: Male subjects able to father children must agree to use two acceptable methods of contraception throughout the study (e.g. condom with spermicidal gel). Double-barrier contraception is required.
8. Negative TB test (e.g. Mantoux or Quantiferon assay).
9. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
10. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures *Women of childbearing potential are defined as females who have experienced menarche, are not postmenopausal (12 months with no menses without an alternative medical cause) and are not permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral oophorectomy or bilateral salpingectomy)

Exclusion Criteria:

1. Second or later glioma progression.
2. Surgical resection or biopsy of glioma within 4 weeks of the start of study treatment.
3. Subjects who participated in an investigational drug or device study within 4 weeks prior to study treatment start.
4. Treatment with tumor-treating fields
5. Radiotherapy within 6 weeks prior to study treatment start.
6. Patients unable to undergo contrast-enhanced MRI.
7. Patient taking herbal medications within 7 days prior to first dose of the study drug.
8. Known history of allergy to TNF, excipient in study medication or any other intravenously administered human proteins/peptides/antibodies.
9. Absolute neutrophil count (ANC) < 1.5 x 10^9/L, platelets < 100 x 10^9/L or haemoglobin (Hb) < 9.0 g/dl.
10. Chronically impaired renal function as indicated by creatinine clearance < 60 mL/min.
11. Inadequate liver function (ALT, AST, ALP ≥ 2.5 x ULN or total bilirubin ≥ 2.0 x ULN)
12. Any severe concomitant condition which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol, in the opinion of the investigator.
13. History within the last year of cerebrovascular disease and/or acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
14. Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria).
15. Clinically significant cardiac arrhythmias or requiring permanent medication.
16. Abnormal LVEF or any other abnormalities observed during baseline ECG and echocardiogram investigations that are considered as clinically significant by the investigator.
17. Uncontrolled hypertension.
18. Ischemic peripheral vascular disease (Grade IIb-IV according to Leriche-Fontaine classification).
19. Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (e.g. risk of doing harm to self or others), or patients with active severe personality disorders.
20. Anxiety ≥ CTCAE grade 3
21. Severe diabetic retinopathy such as severe non-proliferative retinopathy and proliferative retinopathy.
22. Major trauma including major surgery (such as abdominal/cardiac/thoracic surgery) within 4 weeks of administration of study treatment.
23. Pregnancy or breast-feeding.
24. Requirement of chronic administration of high dose corticosteroids or other immunosuppressant drugs. Subjects must have been either off corticosteroids, or on a stable or decreasing dose ≤ 10 mg daily prednisone (or equivalent) for at least 2 weeks prior to study treatment start. Limited or occasional use of corticosteroids to treat or prevent acute adverse reactions is not considered an exclusion criterion.
25. Presence of active and uncontrolled infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
26. Concurrent malignancies, unless the patient has been disease-free for at least 2 years.
27. Growth factors or immunomodulatory agents within 7 days prior to the administration of study treatment.
28. Serious, non-healing wound, ulcer or bone fracture.
29. Requirement of concurrent therapy with anticoagulants at therapeutic doses.
30. Requirement of concurrent use of other anti-cancer treatments or agents other than study medication.
31. Any recent live vaccination within 4 weeks prior to treatment or plan to receive vaccination during the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicity (DLT) | From the first day of treatment until the end of the DLT window (up to 21 days)
Adverse event (AE), Serious Adverse Events (SAE) and Drug Induced Liver Injury (DILI) assessment based on CTCAE v.5.0 | From the inclusion in the study (signature of the informed consent form - ICF) until the end of follow-up (up to approximately 36 months)
Standard laboratory (haematology, biochemistry, liver and urine analysis) parameters | From the inclusion in the study (signature of the informed consent form - ICF) until the end of follow-up (up to approximately 36 months)
Neurological assessment using the Neurologic assessment in Neuro-Oncology (NANO) scale | From the inclusion in the study (signature of the informed consent form - ICF) until the end of follow-up (up to approximately 36 months)
  Measurement of neurological function in neuro-oncology
Karnofsky Performance Status | From the inclusion in the study (signature of the informed consent form - ICF) until the end of follow-up (up to approximately 36 months)
  Assessment through a questionnaire of symptom-related restriction of activity, self-sufficiency and self-determination
Electrocardiogram (ECG) findings. In particular, data about QT/QTc intervals will be collected and analysed for QT/QTc prolongation potentially caused by treatment. | From the inclusion in the study (signature of the informed consent form - ICF) until the end of follow-up (up to approximately 36 months)
Echocardiogram (ECHO) findings. In particular, data about QT/QTc intervals will be collected and analysed for QT/QTc prolongation potentially caused by treatment. | From the inclusion in the study (signature of the informed consent form - ICF) until the end of follow-up (up to approximately 36 months)
Assessment of the formation of human anti-fusion protein antibodies (HAFA) against L19TNF. | Cycle 1 day 1 - First Follow Up visit (up to approximately 9 months)
Progression-free survival (PFS), according to iRANO (immunotherapy response assessment in neuro-oncology) criteria based on standardized MRI protocol | At 6 months

SECONDARY OUTCOMES:
Progression free survival (PFS) | From the inclusion in the study (signature of the informed consent form - ICF) until the end of follow-up (up to approximately 12 months)
Overall survival (OS). | From the inclusion in the study (signature of the informed consent form - ICF) until the end of follow-up (up to approximately 36 months)
Overall Response Rate (ORR, consisting of Complete and partial Response), based on iRANO criteria. | At 12 weeks, 18 weeks, 24 weeks, 36 weeks, 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Weiss, MD, Principal Investigator — Universitätsspital Zürich
Locations (3):
- Switzerland (3):
  - Inselspital Bern, Bern
  - CHUV Départment d'Oncologie, Lausanne
  - Universitatspital Zurich - Klinik fur Neurologie & Hirntumorzentrum, Zurich

IPD SHARING:
Plan to Share IPD: No